CLINICAL TRIAL: NCT02028286
Title: A Phase 1, Open Label, Multiple Center Study to Evaluate the Pharmacokinetics of Once-Daily CLS001 Topical Gel Under Maximal Use Conditions Administered for 21 Days in Subjects With Papulopustular Rosacea
Brief Title: A 21 Day Pharmacokinetics Study in Papulopustular Rosacea
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Maruho Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLS001-CO-PR-002
Record Dates: First submitted 2013-11-27; First posted 2014-01-07 (Estimated); Last update posted 2014-04-14 (Estimated); Status verified 2014-04

CONDITIONS: Papulopustular Rosacea
Keywords: Rosacea
MeSH Terms: conditions — Rosacea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CLS001 (Experimental): CLS001
  Interventions: Drug: CLS001

INTERVENTIONS:
Drug: CLS001

SUMMARY:
The purpose of this study is to characterize the pharmacokinetics of once daily topical gel and confirm that steady state conditions are reached under maximal use conditions following 3 weeks of daily applications.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of papulopustular rosacea
* Grade 3 or 4 on the 5-point Investigator Global Assessment scale
* Presence of telangiectasia

Exclusion Criteria:

* steroid rosacea or subtype 3 (phymatous rosacea)
* clinically significant abnormal findings that would interfere with study objective or risk to safety for the subject.
* nodular rosacea (lesions greater than 5mm with more than 2 modules)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-01; Primary Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Plasma concentrations of CLS001 to determine pharmacokinetic parameters at visit 2, visit 3 and visit 5 | 24 days
  Plasma concentrations of CLS001 to determine pharmacokinetic parameters at visit 2, visit 3 and visit 5.

SECONDARY OUTCOMES:
incidence of adverse events | 24 days

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Frontage Clinical Services, Hackensack, New Jersey
  - Derm Research, Austin, Texas